CLINICAL TRIAL: NCT06621420
Title: Peyronie Disease Questionnaire (PDQ): Turkish Validation
Acronym: Turkish PDQ
Status: Enrolling by invitation | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Burak Citamak, Associate Professor, Acibadem University
Other Study IDs: 2024-8/314
Record Dates: First submitted 2024-09-04; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Peyronie Disease
Keywords: Peyronie; Questionnaire; validation
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the present study is to translate into the Turkish and a perform a validation of the Turkish version of a PDQ and to ensure the use of Turkish validation of the PDQ in clinical use and studies.

DETAILED DESCRIPTION:
The Peyronie Disease Questionnaire (PDQ) The PDQ is a 15-item, self-administered, disease-specific, and multidimensional printed format instrument developed to quantify the psychosexual symptoms of PD. The PDQ includes three scales: ;psychological and physical symptoms; (6 items) ;penile pain; (3 items), and ;symptom bother; (4 scored items and 2 yes/no questions). The ;psychological and physical symptom; domain has a 5-level Likert scale ranging from ;none; to ;very severe.; Patients must complete items on the ;penile pain; domain thinking about the last 24 h, and a numeric scale ranging from 0 to 10 was used to evaluate its severity. The;symptom bother; domain has a 5-level Likert scale (not at all bothered; a little bit bothered, ;moderately bothered,very ;and extremely bothered). The sum of all responses is calculated and given separately for each domain, as long as a total PDQ score is not intended. Higher domain scores indicate a greater negative impact, being the score range from 0 to 24 for ;psychological and physical symptom; from 0 to 30 for ;penile pain and from 0 to 16 for ;symptom bother

The PDQ translation procedure followed a structured method to ensure reliability. The translation method included the following steps: 1. Translation of the original questionnaire to Spanish by two independent professional translators. 2. Merging both translated versions by the research team. 3. Back translation of the merged version by two native English professional translators. 4. Review of the different back-translated English versions with the original questionnaire by the research team. 5. Revising the conceptual equivalence with the original, performed by both the translators and the researchers. 6. Testing the translated questionnaire in a pilot group of 30 patients. 7. Results analysis of the pilot test and completion of translation by the research team. 8. Final editions of the questionnaire. 9. Final report of the researchers.

This study included a total of 60 patients with a diagnosis of PD excluding those who had previously received invasive treatment. Males over 18 years of age and patients diagnosed with Peyronie disease who had not undergone surgery were included in the study.

The test-retest reliability of the PDQ-I and the internal consistency of its subscales will be assessed. Intraclass correlation coefficients (ICC) will be calculated to assess the degree of association between the PDQ subscale scores. Paired Student t-tests will be used to assess whether there are statistically significant score changes between T1 and T2. Internal consistency reliability will be assessed by calculating Cronbachs alpha for each of the three PDQ subscales.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years),
* men,
* diagnosis of PD, except those who have previously received invasive treatment

Exclusion Criteria:

* had an insufficient level of Turkish to write and/or understand the methodology of the questionnaire and follow the guidelines described,
* had previously received an invasive treatment

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Peyronie's disease is a male disease associated with penile deformity, so only male patients were included in the study.
Study Population: Men living in the Marmara region whose native language is Turkish
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Reliability and usability of the Turkish translation of the PDQ | From September 2024 to April 2025
  The scores given by the patients according to the previously proven PDQ scoring will be compared statistically. As a result of this comparison, it will be investigated how consistent and reliable the translation is. The measurement tool in this study is the Peyronie disease questionnaire. The PDQ is a 15-item, self-administered, disease-specific, and multidimensional printed format instrument developed to quantify the psychosexual symptoms of PD. The PDQ includes three scales: "psychological and physical symptoms" (6 items), "penile pain" (3 items), and "symptom bother" (4 scored items and 2 yes/no questions). The "psychological and physical symptom" domain has a 5-level Likert scale ranging from "none" to "very severe." Patients must complete items on the "penile pain" domain thinking about the last 24 h, and a numeric scale ranging from 0 to 10 was used to evaluate its severity. The "symptom bother" domain has a 5-level Likert scale ("not at all bothered," "a little bit bothered,").

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Hellstrom WJ, Feldman R, Rosen RC, Smith T, Kaufman G, Tursi J. Bother and distress associated with Peyronie's disease: validation of the Peyronie's disease questionnaire. J Urol. 2013 Aug;190(2):627-34. doi: 10.1016/j.juro.2013.01.090. Epub 2013 Jan 31. PMID 23376705
- [Background] Garcia-Gomez B, Martinez-Salamanca JI, Sarquella-Geli J, Justo-Quintas J, Garcia-Rojo E, Fernandez-Pascual E, Ruiz-Castane E, Romero-Otero J. Correction: Peyronie's Disease Questionnaire (PDQ): Spanish translation and validation. Int J Impot Res. 2024 Feb;36(1):102. doi: 10.1038/s41443-023-00734-0. No abstract available. PMID 37464022
- [Background] Traunero F, Di Grazia M, Ongaro L, Rizzo M, Cocci A, Verze P, Zucchi A, Cai T, Salame L, Garaffa G, Trombetta C, Liguori G. Validation of the Italian version of the Peyronie's Disease Questionnaire (PDQ). Int J Impot Res. 2024 Sep;36(6):588-591. doi: 10.1038/s41443-023-00792-4. Epub 2023 Nov 17. PMID 37978202